CLINICAL TRIAL: NCT02821442
Title: "Electro Acupuncture in the Treatment and Management of Chemotherapy Induced Peripheral Neuropathy"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: CancerCare Manitoba (Other)
Responsible Party: Principal Investigator, Barbara Shay, Associate Professor, Department head, College of Rehabilitation Sciences, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H2015:282
Record Dates: First submitted 2015-12-08; First posted 2016-07-01 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: Electroacupuncture; Neuropathic Pain; Chemotherapy Induced Peripheral Neuropathy
MeSH Terms: conditions — Breast Neoplasms; Neuralgia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture will consist of acupuncture points ST36, LR3, LI4 bilaterally x 30 minutes, once a week over 6 weeks. ST36 will have EA with 2Hz at the maximum tolerated intensity (ES-130 Portable Japanese Electro-Acupuncture Device, UPC Medical Supplies Inc. South El Monte, CA, USA).
  Interventions: Device: Acupuncture
- Sham Acupuncture (Sham Comparator): Sham acupuncture (Streitberger Placebo Needles, Asiamed) uses the same points and treatment parameters but the placebo needle does not penetrate the skin and the current for EA is not turned on.
  Interventions: Device: Sham Acupuncture

INTERVENTIONS:
Device: Acupuncture — Acupuncture points selected on the arms and legs using both acupuncture and electroacupuncture to assess effectiveness in alleviating neuropathic pain caused by chemotherapy in breast cancer patients
  Arms: Acupuncture
Device: Sham Acupuncture — Placebo needles appear to penetrate but do not actually penetrate the skin
  Arms: Sham Acupuncture

SUMMARY:
To evaluate the effectiveness of Electro acupuncture (EA) for treatment of persistent painful CIPN symptoms in patients with stages 1-3 breast cancer treated with docetaxel chemotherapy 6 months prior

DETAILED DESCRIPTION:
A double blind prospective randomized controlled pilot study with cross over.

To assess the effectiveness of EA in improving pain and function for chronic chemotherapy Induced Peripheral Neuropathy (CIPN) 30 participants will be recruited 6 months post-completion of chemotherapy. Fifteen participants will be randomized to the true EA group and 15 to the sham EA group. Those participants randomized to the sham group will cross over to receive true EA after the trial is complete.

Treatment consists of EA or sham EA 1 x per week x 6 weeks. Re-assessment visits occur after the 6 week intervention and again 2 months post trial.

Each assessment visit quantifies the sensory experience of CIPN at that moment in time using Quantitative Sensory Testing (QST) which includes; thermal detection and thermal pain thresholds, light touch detection using nylon monofilament hairs (Semmes Weinstein Monofilaments (SWMF)), static 2-point discrimination, pressure algometry and vibration thresholds. Patient reported outcome measures including the Disabilities of the Arm, Shoulder and Hand (DASH), Lower extremity functional score (LEFS), the Self report Leeds Assessment of Neuropathic signs and symptoms (S-LANSS) pain questionaire will also be used.

ELIGIBILITY:
Inclusion Criteria:

* Any patient diagnosed with stage 1-3 breast cancer who has finished chemotherapy 6 months prior and has residual CIPN symptoms graded as a 3/10 or higher on the numeric rating pain scale.

Exclusion Criteria:

* Patients who have co-morbid conditions that cause peripheral neuropathic symptoms
* patients with heart valve replacements
* patients on prophylactic antibiotics
* patients with severe coagulopathy
* patients who did not receive regular taxane therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
S-Lanss (short- Leads assessment of neuropathic symptoms and signs) | 2 years
  16 point pain questionnaire that differentiates nociceptive from neuropathic pain
VAS (Visual Analogue Scale) | 2 years
  10 point verbal rating pain scale to measure participants pain in each assessment
DASH (Disabilities of the arm, shoulder, hand) | 2 years
  30 item questionnaire measuring upper limb function
LEFS (Lower extremity functional scale) | 2 years
  20 item questionnaire measuring lower limb function

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Shay, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes